CLINICAL TRIAL: NCT00171184
Title: Efficacy, Safety, and Tolerability of Darifenacin in Patients Aged > 65 Years With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDAR328A2409
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder, Darifenacin, M3 muscarinic receptor antagonist, elderly population
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Darifenacin
  Interventions: Drug: Darifenacin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darifenacin — Darifenacin 7,5 mg tablets once daily with the possibility to up-titrate to 15 mg once daily
  Other Names: Enablex
  Arms: 1
Drug: Placebo — Placebo tablet once daily with sham titration
  Arms: 2

SUMMARY:
The objective of this study is to assess the efficacy, safety and tolerability of 12-weeks treatment with darifenacin in patients aged >Ý 65 years with OAB.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB for at least six months prior to Visit 3
* Symptoms of OAB during the 7 day diary period immediately preceding Visit 3:
* ≥ 1 UUIE on average per day and
* ≥ 10 episodes of micturition on average per day

Exclusion Criteria:

* A total daily urinary volume > 3000 ml or a mean volume voided per micturition of > 300 ml as verified in the micturition diary before randomization
* Post-void residual (PVR) urinary volume > 100 ml
* Clinically significant stress urinary incontinence as determined by the investigator
* Clinically significant bladder outlet obstruction as determined by the investigator
* Concomitant diseases in which the use of anticholinergic drugs is contraindicated, e.g. urinary retention, gastric retention, uncontrolled narrow-angle glaucoma, myasthenia gravis, severe hepatic impairment (Child Pugh B and C), severe ulcerative colitis, toxic megacolon.

Other protocol inclusion / exclusion criteria may apply

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-04; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of urge urinary incontinence episodes (UUIE) per week at week 12.

SECONDARY OUTCOMES:
Change from baseline in : number of UUIE per week at week 1, 2 and 6, number of micturitions per day at week 1,2 and 12; number of urinary incontinence pads used per week at week 1,2,6 & 12; number of nocturnal voids per week at week 1,2,6 & 12.
Safety and tolerability.
Quality of life at week 6 and/or 12.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — East Hanover NJ
Locations (1):
- Scott Department of Urology Baylor College of Medicine, Houston, Texas, United States